CLINICAL TRIAL: NCT02933684
Title: D-Cycloserine and Virtual Reality Exposure Therapy Delivered on an iPad: Increasing Access to Treatment for Social Anxiety Disorder
Brief Title: D-Cycloserine and Virtual Reality Exposure Therapy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to access components necessary to be able to run the study.
Sponsor: Georgia State University (Other)
Collaborators: Emory University (Other)
Responsible Party: Principal Investigator, Page Anderson, Associate Professor, Georgia State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ULTR000454
Record Dates: First submitted 2015-05-05; First posted 2016-10-14 (Estimated); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Social Anxiety Disorder
MeSH Terms: conditions — Phobia, Social | interventions — Cycloserine; Virtual Reality Exposure Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DCS (Experimental): Participants will receive 50mg of Seromycin (aka D-cycloserine) in conjunction with virtual reality exposure therapy once a week for 4 weeks.
  Interventions: Drug: Seromycin; Behavioral: Virtual Reality Exposure Therapy
- Placebo (Placebo Comparator): Participants will receive a placebo in conjunction with virtual reality exposure therapy once a week for 4 weeks.
  Interventions: Behavioral: Virtual Reality Exposure Therapy; Drug: Placebo

INTERVENTIONS:
Drug: Seromycin — Seromycin (aka D-cycloserine) is an analogue of D-alanine and a partial agonist at the NMDA receptor, which facilitates the process of fear extinction.
  Other Names: D-cycloserine
  Arms: DCS
Behavioral: Virtual Reality Exposure Therapy — Allows for delivery of exposure therapy on an iPad. Participants read a speech to a virtual audience. Exposures become increasingly more difficult as the audience becomes more hostile and speeches increase in length and complexity.
Drug: Placebo — Administered in pill form.
  Arms: Placebo

SUMMARY:
The proposed project aims to increase accessibility of exposure therapy, an evidence based treatment for social anxiety disorder, by adapting a therapist-assisted computer-based program to be delivered in a self-guided manner on an iPad. A significant problem with self-guided treatment delivered via computer is compliance. The vast majority of users do not complete treatment, so achieving therapeutic benefit as quickly as possible is essential. D-cycloserine is a drug found to augment response to therapist-guided exposure therapy for anxiety disorders, but has never been tested with self-guided exposure. This study uses a randomized, double-blind methodology to compare D-cycloserine (50 mg; DCS) to placebo in combination with self-guided virtual reality exposure therapy (VRE) delivered via iPad to treat social anxiety disorder. The proposed study tests the hypothesis that patients who receive DCS in combination with the self-guided VRE will show more improvement than those who receive placebo in combination with VRE. Outcome measures include self-reported symptoms of social anxiety, behavioral avoidance, and diagnostic remission. Participants (N=34) are adults with a primary diagnosis of social anxiety disorder. Participants will complete a structured diagnostic interview, standardized self-report measures of social anxiety, and a behavioral avoidance task (i.e., giving a speech) and will be assessed at pre-treatment, at post-treatment and at 3 month follow-up. Hierarchical linear regression and chi-square analyses will be used to test differences between those randomized to DCS versus placebo on the following outcomes: post-treatment scores of self-reported social phobia symptoms, willingness to and anxiety while giving a speech at post-treatment, and diagnostic remission at 3 month follow-up. The proposed project combines technological advances with translational research to develop an innovative and accessible treatment for those with social anxiety disorder. The pilot data generated from this study will be appealing to a variety of funding agencies, including the National Institute of Mental Health's call for exploratory clinical trials of novel interventions for mental illnesses, the Patient-Centered Outcomes Research Institute's call for effectiveness studies aimed to overcome barriers to treatment, and the National Science Foundation's call for innovation-technology translation research.

DETAILED DESCRIPTION:
Social Anxiety Disorder (social phobia) is the most common psychiatric disorder in the US. It negatively impacts health-related quality of life, educational and economic achievement, and it leads to attempted suicide in as many as 21% of affected individuals. A critical barrier to progress in reducing the negative impact of this disorder is that 75-92% of sufferers do not receive treatment. Social phobia self-help programs delivered via computer are designed to increase access to treatment and can be effective. Compliance and completion rates of such programs are, however, quite poor, greatly limiting their impact and accessibility. Furthermore, self-help programs for social phobia do not directly administer a critical component of treatment - exposure therapy. The direct administration of self-guided exposure therapy, using virtual reality is an innovation that would increase the accessibility and impact of computer delivered treatment.

Exposure therapy is based on well-researched fear extinction learning paradigms, where individuals confront what they fear in a therapeutic manner and learn that the feared outcome will not occur. Ressler et al's groundbreaking translational research showed that D-cycolserine (DCS), an analogue of D-alanine and a partial agonist at the NMDA receptor, facilitates the process of fear extinction. DCS is different from other pharmacological agents used to treat social phobia which are prescribed chronically (daily) over a period of months or years to maintain a therapeutic dose; one pill of DCS is taken immediately before exposure therapy sessions. This work sparked a flurry of research showing that DCS augments exposure therapy for a variety of anxiety disorders; people who take DCS show benefit from therapist-assisted exposure therapy more quickly than those who take placebo. Two randomized double-blind, placebo-controlled studies of social phobia conclude that the combination of DCS and therapist-assisted exposure therapy improves treatment response when participants complete fewer exposure sessions. The ability of DCS to speed up the response to exposure therapy is especially valuable for sufferers using self-guided treatment, because they are not generally compliant with the full exposure protocol. The combination of DCS and self-guided exposure therapy would increase access to effective treatment. The use of DCS with self-guided exposure, however, has never been tested.

Specific Aims

1. Adapt an existing computer program to deliver self-guided VRE for social phobia via iPad, and
2. Test the comparative efficacy of DCS vs placebo plus self-guided VRE.

Hypothesis: Participants who receive self-guided VRE plus DCS will show less self-reported social anxiety and less avoidance during a laboratory based behavioral test following a 5-week intervention than those who received self-guided VRE plus placebo.

The investigators seek to shift current clinical practice in the treatment of social phobia so that more people with the disorder receive exposure therapy. The investigators will improve access to evidence-based treatment for social phobia with delivery of exposure via a computer - a modality that capitalizes on the fact that people with severe social phobia spend extensive hours on the computer; exposure therapy can come to people with social phobia "where they are." The investigators also will be the first to test the delivery of exposure therapy on an iPad. The study design improves the approach of existing research on computer-delivered programs for social phobia by testing how treatment affects real behavior - existing research has relied exclusively on self-report measures and assessment of diagnostic status. No studies have assessed actual behavior - either in the lab or in the real-world. This study will improve scientific knowledge by answering the question of whether or not DCS augments self-guided exposure therapy. The combination of a self-help program with DCS addresses many of the obstacles to treatment with therapist-guided exposure therapy. For example, there are not enough mental health providers trained in exposure therapy. Furthermore, social anxiety disorder is characterized by the fear and avoidance of social situations, and psychotherapy is inherently a social encounter. The effective combination of DCS and self-guided virtual reality exposure is an avenue for treatment to any sufferer with access to a computer and a prescribing physician. When the proposed aims are achieved, an innovative treatment will exist that did not before - self-guided VRE delivered via computer.

The investigators have developed and tested a self-help program delivered via computer, with minimal therapist support. The self-help program was tested in a small (N=10) uncontrolled trial of 8 sessions, and results showed decreases in scores on standardized self-report measures of social anxiety from pre- to post-treatment and follow-up. Large effect sizes were observed at post-treatment (d = 1.22-1.53) and follow-up (d = 1.41 - 2.39).

Using standardized measures of software usability, participants described the program as easy-to-use, including a participant who had never before used a computer. Since this study, the program has been updated with new virtual environments, as well as shortening the treatment down. The proposed project will adapt an existing program for delivery via a tablet and to collect data via the computer.

Finally, the investigative team completed a double-blind, placebo controlled trial that tested the combination of DCS vs placebo combined with therapist-guided VRE for specific phobia.

Thus, the investigative team is well-positioned to complete the specific aims of adapting a computer program that delivers self-guided exposure therapy for social phobia via a tablet and testing following hypothesis: Participants who receive self-guided exposure therapy plus DCS will show less self-reported social anxiety and less avoidance during a laboratory based behavioral test following a 5-week intervention than those who received self-guided exposure therapy plus placebo.

ELIGIBILITY:
Inclusion Criteria:

* Understand and provide written informed consent prior to conduct of any study procedures.
* Be able to communicate in English with study personnel
* Be able to manipulate the computer interface to interact with the program
* If female, must have a negative pregnancy test prior to treatment and be maintained on an acceptable method of birth control during treatment
* If using psychotropic medication, stable on medication and dosage for 3 months

Exclusion Criteria:

* Participation in clinical trial within the past 12 months or treatment with DCS in a previous study
* History of mania, schizophrenia, or other psychoses
* Any unstable medical condition; Seizure disorders, with the exception of a childhood history of isolated, non-recurrent febrile seizures
* Current or past substance (except nicotine, caffeine) or alcohol dependence based on DSM-V criteria within six months prior to screening
* Liebowitz Social Anxiety Scale (LSAS) score of < 50 at baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01-01 (Estimated); Primary Completion 2016-12-31 (Estimated); Study Completion 2016-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in scores on the Liebowitz Social Anxiety Scale-self report version (LSAS-SR) | Participants will complete this measure once a week for 6 weeks and again at 17 weeks after the first visit.
  Measures fear in and avoidance of 24 social situations.
Change in behavioral avoidance | Week 1, week 7, and 17 weeks after the first session.
  Complete Unstructured Conversation and Impromptu Speech Tasks. The assessments will be video recorded and the amount of eye contact - in seconds - will be rated by blind observers. The number of seconds of eye contact can then be compared across time points.
Change in scores on the Clinical Global Improvement Scale, Patient Report | Week 7
  Assesses diagnostic remission.

SECONDARY OUTCOMES:
Change in scores on the Social Phobia Scale | Participants will complete this measure once a week for 6 weeks and again at 17 weeks after the first visit.
  Assesses fears of being scrutinized during performance situations.
Change in scores on the Social Interaction Anxiety Scale | Participants will complete this measure once a week for 6 weeks and again at 17 weeks after the first visit.
  Assesses the cognitive, affective, and behavioral reactions to social interactions.
Change in scores on the Patient Health Questionnaire | Week 1, week 7.
  Assesses depressive symptoms.
Change in scores on the Sheehan Disability Scale | Week 1, week 7.
  Assesses functional impairment across work, social life, and family life.
Change in scores on the Quality of Life Inventory | Week 1, week 7.
  Assesses the degree of satisfaction across important life domains.

CONTACTS AND LOCATIONS:
Overall Officials: Page Anderson, PhD, Principal Investigator — Georgia State University
Locations (1):
- Georgia State University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schneier FR, Heckelman LR, Garfinkel R, Campeas R, Fallon BA, Gitow A, Street L, Del Bene D, Liebowitz MR. Functional impairment in social phobia. J Clin Psychiatry. 1994 Aug;55(8):322-31. PMID 8071299
- [Background] Schneier FR, Johnson J, Hornig CD, Liebowitz MR, Weissman MM. Social phobia. Comorbidity and morbidity in an epidemiologic sample. Arch Gen Psychiatry. 1992 Apr;49(4):282-8. doi: 10.1001/archpsyc.1992.01820040034004. PMID 1558462
- [Background] Andrews G, Cuijpers P, Craske MG, McEvoy P, Titov N. Computer therapy for the anxiety and depressive disorders is effective, acceptable and practical health care: a meta-analysis. PLoS One. 2010 Oct 13;5(10):e13196. doi: 10.1371/journal.pone.0013196. PMID 20967242
- [Background] Christensen H, Griffiths KM, Jorm AF. Delivering interventions for depression by using the internet: randomised controlled trial. BMJ. 2004 Jan 31;328(7434):265. doi: 10.1136/bmj.37945.566632.EE. Epub 2004 Jan 23. PMID 14742346
- [Background] Kroenke K, Spitzer RL, Williams JB, Monahan PO, Lowe B. Anxiety disorders in primary care: prevalence, impairment, comorbidity, and detection. Ann Intern Med. 2007 Mar 6;146(5):317-25. doi: 10.7326/0003-4819-146-5-200703060-00004. PMID 17339617
- [Background] Hofmann SG, Sawyer AT, Asnaani A. D-cycloserine as an augmentation strategy for cognitive behavioral therapy for anxiety disorders: an update. Curr Pharm Des. 2012;18(35):5659-62. doi: 10.2174/138161212803530916. PMID 22632472
- [Background] Hofmann SG, Meuret AE, Smits JA, Simon NM, Pollack MH, Eisenmenger K, Shiekh M, Otto MW. Augmentation of exposure therapy with D-cycloserine for social anxiety disorder. Arch Gen Psychiatry. 2006 Mar;63(3):298-304. doi: 10.1001/archpsyc.63.3.298. PMID 16520435
- [Background] Guastella AJ, Richardson R, Lovibond PF, Rapee RM, Gaston JE, Mitchell P, Dadds MR. A randomized controlled trial of D-cycloserine enhancement of exposure therapy for social anxiety disorder. Biol Psychiatry. 2008 Mar 15;63(6):544-9. doi: 10.1016/j.biopsych.2007.11.011. Epub 2008 Jan 7. PMID 18179785
- [Background] Caplan SE. Relations among loneliness, social anxiety, and problematic Internet use. Cyberpsychol Behav. 2007 Apr;10(2):234-42. doi: 10.1089/cpb.2006.9963. PMID 17474841
- [Background] Anderson PL, Price M, Edwards SM, Obasaju MA, Schmertz SK, Zimand E, Calamaras MR. Virtual reality exposure therapy for social anxiety disorder: a randomized controlled trial. J Consult Clin Psychol. 2013 Oct;81(5):751-60. doi: 10.1037/a0033559. Epub 2013 Jun 24. PMID 23796315
- [Background] Anderson P, Zimand E, Schmertz SK, Ferrer M. Usability and utility of a computerized cognitive-behavioral self-help program for public speaking anxiety. Cognitive and Behavioral Practice 14(2):198-207. 2007.
- [Background] Ressler KJ, Rothbaum BO, Tannenbaum L, Anderson P, Graap K, Zimand E, Hodges L, Davis M. Cognitive enhancers as adjuncts to psychotherapy: use of D-cycloserine in phobic individuals to facilitate extinction of fear. Arch Gen Psychiatry. 2004 Nov;61(11):1136-44. doi: 10.1001/archpsyc.61.11.1136. PMID 15520361
- [Background] Heimberg RG, Horner KJ, Juster HR, Safren SA, Brown EJ, Schneier FR, Liebowitz MR. Psychometric properties of the Liebowitz Social Anxiety Scale. Psychol Med. 1999 Jan;29(1):199-212. doi: 10.1017/s0033291798007879. PMID 10077308
- [Background] Safren SA, Heimberg RG, Horner KJ, Juster HR, Schneier FR, Liebowitz MR. Factor structure of social fears: The Liebowitz Social Anxiety Scale. J Anxiety Disord. 1999 May-Jun;13(3):253-70. doi: 10.1016/s0887-6185(99)00003-1. PMID 10372341
- [Background] Mattick RP, Clarke JC. Development and validation of measures of social phobia scrutiny fear and social interaction anxiety. Behav Res Ther. 1998 Apr;36(4):455-70. doi: 10.1016/s0005-7967(97)10031-6. PMID 9670605
- [Background] Spitzer RL, Kroenke K, Williams JB. Validation and utility of a self-report version of PRIME-MD: the PHQ primary care study. Primary Care Evaluation of Mental Disorders. Patient Health Questionnaire. JAMA. 1999 Nov 10;282(18):1737-44. doi: 10.1001/jama.282.18.1737. PMID 10568646
- [Background] Kadouri A, Corruble E, Falissard B. The improved Clinical Global Impression Scale (iCGI): development and validation in depression. BMC Psychiatry. 2007 Feb 6;7:7. doi: 10.1186/1471-244X-7-7. PMID 17284321
- [Background] Turner SM, Beidel DC, Cooley MR, Woody SR, Messer SC. A multicomponent behavioral treatment for social phobia: social effectiveness therapy. Behav Res Ther. 1994 May;32(4):381-90. doi: 10.1016/0005-7967(94)90001-9. PMID 8192637
- [Background] Beidel DC, Turner SM, Jacob RG, Cooley MR. Assessment of social phobia: Reliability of an impromptu speech task. Journal of Anxiety Disorders 3(3):149-158. 1989.
- [Background] Deveney CM, McHugh RK, Tolin DF, Pollack MH, Otto MW. Combining D-cycloserine and exposure-based CBT for the anxiety disorders. Clin Neuropsychiatry 6(2):75-82. 2009.
- [Background] Hofmann SG. Enhancing exposure-based therapy from a translational research perspective. Behav Res Ther. 2007 Sep;45(9):1987-2001. doi: 10.1016/j.brat.2007.06.006. Epub 2007 Jun 17. PMID 17659253